CLINICAL TRIAL: NCT05063929
Title: An Investigation of the Impact of Fruit on the Gut Microbiota and Its Metabolites: Connections to Human Health
Brief Title: Impacts of Fruit on the Gut Health and Human Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Shirin Hooshmand, Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5A297A
Record Dates: First submitted 2021-02-25; First posted 2021-10-01 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Cardiometabolic Health; Healthy Aging; Cognition
Keywords: Metabolome; Microbiome; Cognition; Fruit intake
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fruits (Experimental): Participants will receive 2 cup eq fruits per day
  Interventions: Other: Fruit (2 cup eq)
- Fruit restriction (Other): Participants will receive 1/2 cup eq fruits per day
  Interventions: Other: Fruit restriction (1/2 cup eq)

INTERVENTIONS:
Other: Fruit (2 cup eq) — participants will receive 2 cup eq fruits
  Arms: Fruits
Other: Fruit restriction (1/2 cup eq) — participants will receive 1/2 cups eq fruits
  Arms: Fruit restriction

SUMMARY:
The objectives of this study are to investigate the effect of fruit consumption on the gut microbiota and their collective fecal and plasma metabolomes, vascular and cardiometabolic functions, cognition, and motor control.

DETAILED DESCRIPTION:
The Investigators findings will provide data critical to the understanding of the effects of fruit intake on the gut microbiome and the capacity of the microbiota to biotransform nutrients contained within fruits as well as the subsequent impact on circulating status of those metabolites. Concurrently, health outcomes that may be linked to these changes including cognition, motor control, vascular function and cardiometabolic health risk markers will be assessed in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women 30 to 70 years old

Exclusion Criteria:

* History of:

  * stroke or myocardial infarction
  * gastrointestinal disorders
  * neurological disorders (epilepsy, multiple sclerosis, Parkinson's disease, stroke, etc)
  * known metabolic disorders (liver, renal or clinically diagnosed diabetes)
  * drug treatment for lipid reduction or hypertension,
  * psychiatric medication use

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in composition of bacterial fecal microbiome at 8 weeks | At baseline, at 8 weeks
  Bacterial fecal microbiome 16S rRNA gene amplicon libraries will be sequence using the Illumina MiSeq next generation sequencing platform.

SECONDARY OUTCOMES:
Change from baseline in processing speed (cognition) at 8 weeks | At baseline, at 8 weeks
  using Pattern Comparison Processing Speed Test
Change from baseline in Vascular health at 8 weeks | At baseline, at 8 weeks
  To better understand how changes in the gut microbiota through fruit consumption are linked to changes in health outcomes, we will assess endothelial function via flow-mediated vasodilation and risk factors for cardiometabolic dysfunction in fasting blood samples collected at baseline and after 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirin Hooshmand, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zingales S, Martinez J, Stepp AH, Miller C, Jason N, Hong MY, Liu C, Kern M, Hooshmand S. Daily Intake of Recommended Servings of Fruit Improves Nutrient Intake but Shows no Major - Effect on Cardiovascular Health or Cognition in Low Fruit Consumers. Curr Dev Nutr. 2025 Sep 3;9(10):107544. doi: 10.1016/j.cdnut.2025.107544. eCollection 2025 Oct. PMID 41081007